CLINICAL TRIAL: NCT02700425
Title: His Bundle Pacing Versus Coronary Sinus Pacing for Cardiac Resynchronization Therapy
Acronym: His-SYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of California, Los Angeles (Other); Northwestern University (Other); Rush University Medical Center (Other); Geisinger Clinic (Other); Indiana University (Other); Edward Hospital (Other); Baptist Health, Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB15-1728
Record Dates: First submitted 2016-01-29; First posted 2016-03-07 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Congestive Heart Failure
Keywords: Wide QRS; Ventricular Dyssynchrony
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- His Bundle Pacing (Active Comparator): Subjects will be randomized to the HB lead position with their cardiac resynchronization therapy (CRT) pacemaker. HB lead pacing will be performed with the Medtronic SelectSecure™, Model 3830 lead. Delivery of the lead utilizes a deflectable sheath, the Medtronic SelectSite™, Model C304. Both devices are FDA approved for the purpose of HB pacing. It is the only device available which is presently FDA approved for selective HB pacing.
  Interventions: Device: CRT Pacemaker
- Coronary Sinus Pacing (Active Comparator): Subjects will be randomized to the CS lead position with their cardiac resynchronization therapy (CRT) pacemaker. CS lead and CRT device generator selected for implant will be left to the discretion of the operator. Only FDA approved CS leads and CRT generators will be utilized in the study. There are five present manufacturers of CS leads and CRT generators: Biotronik, Boston Scientific, Medtronic, Sorin, and St. Jude Medical.
  Interventions: Device: CRT Pacemaker

INTERVENTIONS:
Device: CRT Pacemaker — Cardiac Resynchronization Therapy (CRT) is the use of a pacemaker with two endocardial leads placed in the right atrium (RA) and right ventricle (RV). The third lead is traditionally placed in a tributary of the coronary sinus (CS) overlying the epicardial surface of the left ventricle (LV). Alternatively, the third lead may be positioned based on mapping of the common His bundle and actively fixed to achieve QRS normalization via direct His bundle capture.

SUMMARY:
The goal of this study is to compare the effectiveness of pacing from a physiologic His bundle (HB) lead position versus with the standard coronary sinus (CS) lead position in subjects with heart failure undergoing cardiac resynchronization therapy (CRT). While placement of left ventricular leads via the coronary sinus has anatomic limitations, we hypothesis that the achievement of QRS narrowing with His bundle capture will be superior for improving systolic function by echocardiographic indices (ejection fraction and strain) and quality of life and decreased rehospitalization and mortality.

DETAILED DESCRIPTION:
This is a randomized, single-blinded study of 40 patients to a strategy of HB pacing versus CS pacing, and remain blinded to their treatment allocation. Both treatment options use standard-of-care, FDA-approved devices. The distinction is only in the allocation toward HB pacing and CS pacing. Treating physicians will be aware of assignment in order to facilitate routine device follow-up. Echocardiographic and electrocardiographic evaluation will also be performed in a blinded manner.

Cross-over is permitted between treatment group allocation if:

* CS lead cannot be placed due to difficult cannulation of the CS, limited branches at the posterolateral or lateral wall, or phrenic nerve capture. These subjects may then cross-over to HB pacing.
* HB pacing subjects may cross-over if HB lead cannot be positioned with adequate stability and reasonable pacing output, or if QRS width does not narrow by at least 20% or to a QRS width of ≤ 130 msec.

Implant procedure will be per routine percutaneous access, as is standard for pacemaker and ICDs. All subjects will receive an FDA-approved cardiac resynchronization therapy pacemaker or defibrillator device, as per standard of care outlined for the subject. In order to facilitate optimal lead placement, arterial access for levo-phase CS angiography and/or LV septal mapping to characterize site of bundle-branch block may also be performed, at the discretion of the implanting physician per his/her standard practice.

Follow-up will be performed at 2 weeks post-implant for incision check and device interrogation as is standard of care. In addition, routine device and clinical follow-up will be scheduled at 1, 3, 6, and 12 months. Electrocardiography (ECG) will be performed pre-implant, prior to hospital discharge, at 3 months, 6 months, and 12 months. Echocardiography will be performed pre-implant and 6 months to evaluate for change in LVEF, chamber dimension, and wall motion with strain imaging as is standard of care in the treatment of patients with advanced heart failure. NYHA functional class and quality of life (utilizing the Kansas City Cardiomyopathy Questionnaire) will be assessed pre-implant and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* LV systolic dysfunction with LVEF ≤ 35%
* Evidence of intraventricular conduction delay with QRS duration > 120 msec
* NYHA Class II, III, and ambulatory Class IV heart failure with either ischemic or nonischemic cardiomyopathy and patients with NYHA Class I symptoms and ischemic cardiomyopathy
* Left ventricular ejection fraction (LVEF) ≤ 35%, sinus rhythm (SR), left bundle-branch block (LBBB) morphology, and QRS duration ≥ 150 msec, and NYHA Class II, III, or ambulatory Class IV patients on goal-directed medical therapy (GDMT) [Class I]
* LVEF ≤ 35%, SR with LBBB with QRS 120-149 msec on GDMT [Class IIa]
* LVEF ≤ 35%, SR with non-LBBB with QRS ≥ 150 msec on GDMT [Class IIa]
* LVEF ≤ 35%, in AF if medication or AV nodal ablation will allow near 100% pacing [Class IIa]
* LVEF ≤ 35% undergoing new or replacement device with anticipated >40% ventricular pacing on GDMT [Class IIa]
* LVEF ≤ 30%, ischemic etiology of HF, SR with LBBB ≥ 150 msec and NYHA Class I symptoms on GDMT [Class IIb]
* LVEF ≤ 35%, SR with non-LBBB with QRS 120-149 msec, NYHA Class III/ambulatory Class IV HF on GDMT [Class IIb] LVEF ≤ 35%, SR with non-LBBB with QRS ≥ 150 msec, NYHA Class II HF on GDMT [Class IIb]

Exclusion Criteria:

* Existing CRT device
* Inability of patient capacity to provide consent for themselves either due to medical or psychiatric comorbidity
* Pregnancy
* Participation in other trials
* Difficulty with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Tung, MD, Principal Investigator — University of Chicago; Gaurav A. Upadhyay, MD, Principal Investigator — University of Chicago
Locations (8):
- United States (8):
  - The University of California, Los Angeles, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Edward Hospital, Naperville, Illinois
  - Indiana University, Indianapolis, Indiana
  - Baptist Health Louisville, Louisville, Kentucky
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Upadhyay GA, Vijayaraman P, Nayak HM, Verma N, Dandamudi G, Sharma PS, Saleem M, Mandrola J, Genovese D, Tung R; His-SYNC Investigators. His Corrective Pacing or Biventricular Pacing for Cardiac Resynchronization in Heart Failure. J Am Coll Cardiol. 2019 Jul 9;74(1):157-159. doi: 10.1016/j.jacc.2019.04.026. Epub 2019 May 9. No abstract available. PMID 31078637
- [Result] Upadhyay GA, Vijayaraman P, Nayak HM, Verma N, Dandamudi G, Sharma PS, Saleem M, Mandrola J, Genovese D, Oren JW, Subzposh FA, Aziz Z, Beaser A, Shatz D, Besser S, Lang RM, Trohman RG, Knight BP, Tung R; His-SYNC Investigators. On-treatment comparison between corrective His bundle pacing and biventricular pacing for cardiac resynchronization: A secondary analysis of the His-SYNC Pilot Trial. Heart Rhythm. 2019 Dec;16(12):1797-1807. doi: 10.1016/j.hrthm.2019.05.009. Epub 2019 May 13. PMID 31096064

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
Started | 21 | 20
Completed | 21 | 19 (1 patient withdrew after randomization)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: All analyses shown are intention-to-treat. Of note, 5 patients from Coronary Sinus Pacing crossed over to His Bundle Pacing, but were analyzed Coronary Sinus Pacing. Likewise, 10 patients from His Bundle Pacing crossed over to the Coronary Sinus Pacing, but they were analyzed as His Bundle Pacing under intention-to-treat analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (11.4) | 63.8 (14.1) | 64.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 14 | 11 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 12 | 25
  African-American | 7 | 5 | 12
  Hispanic | 1 | 1 | 2
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40
Height [Mean (Standard Deviation); unit: cm] | 172.4 (9.6) | 166.5 (13.3) | 169.6 (11.7)
Weight [Median (Inter-Quartile Range); unit: kg] | 88.0 [80.9 to 93.0] | 78.0 [64.0 to 89.0] | 83.5 [77.1 to 91.0]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 29.4 [26.1 to 31.3] | 29.4 [26.4 to 32.8] | 29.4 [26.3 to 32.1]
Hypertension (HTN) [Count of Participants; unit: Participants]
  Hypertension | 16 | 14 | 30
  No Hypertension | 5 | 5 | 10
Coronary Artery Disease (CAD) [Count of Participants; unit: Participants]
  CAD | 13 | 13 | 26
  No CAD | 8 | 6 | 14
History of Coronary-Artery Bypass Graft (CABG) [Count of Participants; unit: Participants]
  CABG | 5 | 2 | 7
  No CABG | 16 | 17 | 33
History of Atrial Fibrillation (AF) [Count of Participants; unit: Participants]
  AF | 8 | 5 | 13
  No AF | 13 | 14 | 27
Chronic Obstructive Pulmonary Disease (COPD) [Count of Participants; unit: Participants]
  COPD | 4 | 6 | 10
  No COPD | 17 | 13 | 30
Diabetes Mellitus Type 2 (DM2) [Count of Participants; unit: Participants]
  DM | 11 | 8 | 19
  No DM | 10 | 11 | 21
Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants]
  CKD | 10 | 9 | 19
  No CKD | 11 | 10 | 21
End-Stage Renal Disease (ESRD) [Count of Participants; unit: Participants]
  ESRD | 1 | 2 | 3
  No ESRD | 19 | 17 | 36
  Unknown | 1 | 0 | 1
New York Heart Association (NYHA) Class [Median (Inter-Quartile Range); unit: stages] — NYHA class determines the functional status of the patient. There are classes I-IV. Class I is no symptoms or limitation of physical activity, II is slight limitation of physical activity but comfortable at rest, III marked limitation of physical activity, and IV is unable to carry any physical activity without discomfort, heart failure symptoms at rest, and discomfort increases with any physical activity as described the American Heart Association (AHA).
  stages | 3.0 [2.5 to 3.0] | 2.5 [2.0 to 3.0] | 3.0 [2.25 to 3.0]
Beta-blocker (BB) [Count of Participants; unit: Participants]
  BB | 21 | 18 | 39
  No BB | 0 | 1 | 1
Angiotensin-converting enzyme inhibitor (ACE-I) [Count of Participants; unit: Participants]
  ACE-I | 5 | 6 | 11
  No ACE-I | 16 | 13 | 29
Angiotensin II Receptor Blocker (ARB) [Count of Participants; unit: Participants]
  ARB | 5 | 5 | 10
  No ARB | 16 | 14 | 30
Angiotensin II Recptor Blocker (ARB)/neprilysin inhibitor [Count of Participants; unit: Participants]
  ARB/neprilysin inhibitor | 5 | 4 | 9
  No ARB/neprilysin inhibitor | 16 | 15 | 31
Amiodarone [Count of Participants; unit: Participants]
  Amiodarone | 4 | 4 | 8
  No Amiodarone | 17 | 15 | 32
Digoxin [Count of Participants; unit: Participants]
  Digoxin | 2 | 4 | 6
  No Digoxin | 19 | 15 | 34
Spironolactone [Count of Participants; unit: Participants]
  Spironolactone | 7 | 7 | 14
  No Spironolactone | 14 | 12 | 26
PR interval (PR) [Median (Inter-Quartile Range); unit: ms] | 186 [170 to 216] | 184 [161 to 205] | 186 [166 to 216]
QRS interval (QRS) [Mean (Standard Deviation); unit: seconds] | 172 (16) | 165 (18) | 168 (18)
QTc [Mean (Standard Deviation); unit: ms] | 484 (48) | 478 (35) | 481 (42)
Left Ventricular end-diastolic volume (LVEDV) [Median (Inter-Quartile Range); unit: mL] | 220 [176 to 304] | 190 [154 to 235] | 201 [163 to 262]
Left Ventricular End-Systolic Volume (LVESV) [Median (Inter-Quartile Range); unit: mL] | 165 [132 to 239] | 126 [104 to 163] | 148 [113 to 186]
Left Ventricular Ejection Fraction (LVEF) [Median (Inter-Quartile Range); unit: percent of ejection fraction] | 26.3 [21.3 to 28.3] | 30.5 [27.1 to 33.9] | 27.8 [23.6 to 31.4]

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular Ejection Fraction (LVEF)
Description: Change in left ventricular ejection fraction (LVEF) as measured by echocardiography in a blinded core lab.
Time Frame: baseline and 6 months
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: ejection fraction percentage
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
Number analyzed (Participants) | 21 | 19
ejection fraction percentage
  Baseline | 26.3 [21.3 to 28.3] | 30.5 [27.1 to 33.9]
  6-months | 31.9 [30.8 to 40.1] | 34.0 [31.6 to 42.1]
Statistical Analysis 1: Comparison: Coronary Sinus Pacing; The sample size was estimated based on the primary endpoint of echocardiographic response to test the hypothesis that an absolute 10% greater improvement in LVEF would be observed with His Bundle Pacing compared to Coronary Sinus Pacing, with a significance level of 0.05 and a power of 0.80. Primary outcome was presented at baseline and 6-months as median (interquartile range) based upon the Shapiro-Wilks test of normality, and then analyzed with the Wilcoxon signed rank test; Test type: Other; p < 0.001, Sign test — P-value was not adjusted for multiple comparisons. Test was two-tailed, considered statistically significant with a p-value <0.05, and conducted using SAS version 9.4 (SAS Institute Inc, Cary, NC) and STATA MP version 15 (College Station, TX); Wilcoxon signed rank test
Statistical Analysis 2: Comparison: His Bundle Pacing; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Sign test — [p-value comment as in outcome 1, analysis 1]; Wilcoxon signed rank test

2. Primary Outcome: Change in QRS Duration
Description: Change in QRS duration as measured by electrocardiography
Time Frame: baseline and 12 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
Number analyzed (Participants) | 21 | 19
ms
  Baseline | 172 (16) | 165 (19)
  1-year | 144 (30) | 152 (30)
Statistical Analysis 1: Comparison: Coronary Sinus Pacing; Primary outcome was presented at baseline and 1-year as means +/- standard deviations based upon the Shapiro-Wilks test of normality, and then analyzed with paired t-tests; Test type: Other — paired t-test; p = 0.002, t-test, 2 sided — P-values are not adjusted for multiple comparisons. Tests were two-tailed, considered statistically significant with a p-value <0.05, and conducted using STATA MP version 15 (College Station, TX)
Statistical Analysis 2: Comparison: His Bundle Pacing; Primary outcome of His Bundle Pacing was presented at baseline and 1-year as means +/- standard deviations based upon the Shapiro-Wilks test of normality, and then analyzed with paired t-tests; Test type: Other — paired t-test; p = 0.002, t-test, 2 sided

3. Primary Outcome: Time to First Cardiovascular Hospitalization or Death
Description: Time to first cardiovascular hospitalization or death in months
Time Frame: Through study completion, an average of 12 months.
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
Number analyzed (Participants) | 21 | 19
months | 10.63 [8.47 to 12] | 11.58 [8.3 to 12]
Statistical Analysis 1: Comparison: His Bundle Pacing vs Coronary Sinus Pacing; Primary outcome of time to first cardiovascular hospitalization or death by His Bundle Pacing compared to Coronary Sinus Pacing presented median and interquartile range in years based upon the Shapiro-Wilks test of normality, and then analyzed with a log rank test; Test type: Other — Log rank test of a survival analysis; p = 0.62, Log Rank — P-value did not need to be adjusted for multiple comparisons. Tests were two-tailed, considered statistically significant with a p-value <0.05, and conducted using STATA MP version 15 (College Station, TX)

4. Secondary Outcome: New York Heart Association (NYHA) Functional Class Change
Description: New York Heart Association (NYHA) functional class change for baseline, 6 months, and 12 months. NYHA class determines the functional status of the patient. There are classes I-IV. Class I is no symptoms or limitation of physical activity, II is slight limitation of physical activity but comfortable at rest, III marked limitation of physical activity, and IV is unable to carry any physical activity without discomfort, heart failure symptoms at rest, and discomfort increases with any physical activity as described the American Heart Association (AHA).
Time Frame: baseline, 6 months, and 12 months
Population: All analyses shown are intention-to-treat. Of note, 5 patients from Coronary Sinus Pacing crossed over to His Bundle Pacing, but were analyzed Coronary Sinus Pacing. Likewise, 10 patients from His Bundle Pacing crossed over to the Coronary Sinus Pacing, but they were analyzed as His Bundle Pacing under intention-to-treat analysis. NYHA class determines the functional status of the patient. There are classes I-IV. Class I is no symptoms and IV is symptoms at rest.
Measure: Median (Inter-Quartile Range); unit: class grade
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
Number analyzed (Participants) | 21 | 19
class grade
  Baseline | 3.0 [2.5 to 3.0] | 2.5 [2.0 to 3.0]
  6-Months: number analyzed (Participants) | 21 | 17
  6-Months | 2.0 [2.0 to 2.5] | 2.0 [1.0 to 2.0]
  1-Year: number analyzed (Participants) | 10 | 7
  1-Year | 3.0 [2.0 to 3.0] | 2.0 [1.0 to 2.0]
Statistical Analysis 1: Comparison: Coronary Sinus Pacing; NYHA functional class of Coronary Sinus Pacing arm was presented at baseline as medians (interquartile ranges) based upon the Shapiro-Wilks test of normality, and then analyzed with a Wilcoxon sign rank test; Test type: Other; p = 0.09, Sign test — [p-value comment as in outcome 2, analysis 1]; Wilcoxon sign rank test
Statistical Analysis 2: Comparison: His Bundle Pacing; NYHA functional class of the His Bundle Pacing arm was presented at baseline and 12 months as medians (interquartile ranges) based upon the Shapiro-Wilks test of normality, and then analyzed with Wilcoxon sign rank test; Test type: Other; p = 0.32, Sign test — [p-value comment as in outcome 2, analysis 1]; Wilcoxon sign rank test

5. Secondary Outcome: Quality of Life Change by Kansas City Questionnaire (KCCQ)
Description: Quality of life change as measured by Kansas City Questionnaire (KCCQ) is a 23-item instrument that is self-administered. KCCQ measures physical function, symptoms (specifically frequency, severity, and recent change), social function, self-efficacy and knowledge, and quality of life. Subscales and Total Score range from minimum of 0-100 (maximum); higher scores show better health status. Developed and validated by Dr. John Spertus,MD of University of Missouri-Kansas City.
Time Frame: baseline and 12 months
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
Number analyzed (Participants) | 21 | 19
score on a scale
  Baseline: number analyzed (Participants) | 18 | 19
  Baseline | 65 [37 to 86] | 70 [42 to 83]
  1-Year: number analyzed (Participants) | 7 | 9
  1-Year | 44 [40 to 93] | 85 [82 to 93]
Statistical Analysis 1: Comparison: His Bundle Pacing; Quality of Life was presented at baseline and 1-year as medians (interquartile range) for patients with His Bundle Pacing based upon the Shapiro-Wilks test of normality, and then analyzed with Wilcoxon signed-rank test; Test type: Other; p = 0.35, Sign test — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Coronary Sinus Pacing; Quality of Life was presented at baseline and 1-year as medians (interquartile range) for patients with Coronary Sinus Pacing based upon the Shapiro-Wilks test of normality, and then analyzed with Wilcoxon signed-rank test; Test type: Other; p = 0.07, Sign test — [p-value comment as in outcome 2, analysis 1]

6. Secondary Outcome: Time to First Cardiovascular Rehospitalization
Description: Time to first cardiovascular rehospitalization in 12 months
Time Frame: Through study completion, an average of 12 months
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
Number analyzed (Participants) | 21 | 19
months | 10.63 [8.47 to 12] | 11.58 [8.3 to 12]
Statistical Analysis 1: Comparison: His Bundle Pacing vs Coronary Sinus Pacing; Primary outcome of time to first cardiovascular rehospitalization by His Bundle Pacing compared to Coronary Sinus Pacing presented median and interquartile range in years based upon the Shapiro-Wilks test of normality, and then analyzed with a log rank test; Test type: Other — Log rank test of a survival analysis; p = 0.14, Log Rank — [p-value comment as in outcome 3, analysis 1]

7. Secondary Outcome: Time to First Treated Ventricular Arrhythmia/Ventricular Tachycardia (VT/VF)
Description: Time to first treated ventricular arrhythmia/ventricular tachycardia (VT/VF) in 12 months
Time Frame: Through study completion, an average of 12 months
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
Number analyzed (Participants) | 21 | 19
months | 10.63 [8.57 to 12] | 11.58 [6.97 to 12]
Statistical Analysis 1: Comparison: His Bundle Pacing vs Coronary Sinus Pacing; Primary outcome of time to first treated VT/VF by His Bundle Pacing compared to Coronary Sinus Pacing presented median and interquartile range in years based upon the Shapiro-Wilks test of normality, and then analyzed with a log rank test; Test type: Other — Log rank test of a survival analysis; p = 0.14, Log Rank — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 1 year.
Description: Adverse events were required to be systematically reported into REDCap at time of procedure.
Arm/Group | His Bundle Pacing | Coronary Sinus Pacing
All-Cause Mortality (participants affected / at risk) | 1/21 | 1/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/24
Other Adverse Events (participants affected / at risk) | 1/21 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | His Bundle Pacing (N=21) | Coronary Sinus Pacing (N=19)
Transient ischemic attack with aphasia (Nervous system disorders) | 0 (0) | 1 (1)
atrial lead microdislodgment (Surgical and medical procedures) | 0 (0) | 2 (2)
hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This pilot study was underpowered to detect differences less than 10% between groups.The criteria for LBBB definitions impact the outcomes of CRT studies. More precise electrophysiologic definitions are necessary to refine patient selection for His bundle pacing. Longer helices, deflectable sheaths with septal orientation and variable curves may further improve His correction rates and stability of thresholds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT02700425/Prot_SAP_000.pdf